CLINICAL TRIAL: NCT04294615
Title: Clinical Response and Safety Following Fecal Microbiota Transplantation by Automatic Methods in Patients With Moderate-Severe Active Ulcerative Colitis
Brief Title: Clinical Response and Safety Following FMT for UC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yujie Zhang, Xijing Hospital of Digestive Diseases, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LL-KY-20150305
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Inflammatory Bowel Diseases; Fecal Microbiota Transplantation
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT through a naso-jejunal tube (Experimental): The purified fecal microbiota was delivered into the intestine through a naso-jejunal tube.
  Interventions: Other: FMT through a naso-jejunal tube
- FMT through TET (Active Comparator): The purified fecal microbiota was delivered into the intestine through a transendoscopic enteral tubing (TET) which is fixed to the cecum with clips under endoscopic guidance.
  Interventions: Other: FMT through TET

INTERVENTIONS:
Other: FMT through a naso-jejunal tube — Prepared feces by automatic methods, then the purified fecal microbiota was delivered into the intestine through a naso-jejunal tube.
  Arms: FMT through a naso-jejunal tube
Other: FMT through TET — Prepared feces by automatic methods, then the purified fecal microbiota was delivered into the intestine through a transendoscopic enteral tubing (TET) which is fixed to the cecum with clips under endoscopic guidance.
  Arms: FMT through TET

SUMMARY:
The study aims to evaluate the clinical efficacy and safety of fecal microbiota transplantation by automatic methods in the treatment of moderate to severe active ulcerative colitis. There are two groups according to FMT pathway ( through a naso-jejunal tube or transendoscopic enteral tubing). Patients were followed up until 2 weeks after the final FMT in hospital.

ELIGIBILITY:
Inclusion Criteria:

- Eligible patients required a diagnosis of ulcerative colitis made by a primary gastroenterologist based upon history, physical exam, laboratory/radiological studies and gastrointestinal histology. All patients were age ≥ 18 year old at the time of enrollment. They had moderate to severe symptoms with a mayo score between 6~12 and an endoscopic subscore ≥2. Patient medication for UC could not have changed for at least one month prior to FMT.

Exclusion Criteria:

- Active or history of intraabdominal abscess, acute abdomen or other clinical emergencies requiring emergent management, pregnancy, prior history of FMT, prior history of TNF inhibitors use, or other serious systemic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
clinical response | 2 weeks after FMT
  reduction in the Mayo score of ≥3 points and ≥30% from baseline, with a decrease in the rectal bleeding subscore of ≥1 point or a subscore of ≤1

SECONDARY OUTCOMES:
clinical remission, safety and progression of disease | 2 weeks after FMT
  clinical remission: Mayo score ≤ 2, with no subscore > 1; progression of disease: measured by initiation of anti-TNFα or colectomy. Adverse event severity and relatedness was graded using NIH criteria.

IPD SHARING:
Plan to Share IPD: No